CLINICAL TRIAL: NCT05722509
Title: Evaluation of a Periodontal Pocket Reduction Technique Applied to Exodontia of Erupted or Semi-erupted Wisdom Teeth
Brief Title: Evaluation of a New Technique for Periodontal Pocket Reduction in the Extraction of Wisdom Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Rosario María Ramírez Puerta, Clinical Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRF1
Record Dates: First submitted 2023-01-20; First posted 2023-02-10 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Molar, Third; Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pre-measurements will be performed by 2 previously calibrated examiners (R.R.P and J.R.M). The calibration will consist of evaluating the periodontal probing of 10 patients in the mesial, distal, vestibular, and palatal/lingual areas and comparing the results of both examiners until an excellent degree of agreement is achieved. The surgical procedure will be performed by the principal investigator (RRM). Measurements of the results in the different study periods will be performed by a third independent evaluator (JFF) who will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Distal Reduction Flap" Group (Experimental): A surgical procedure consisting of a tissue reduction flap distal to the second molar prior to the extraction of the third molar will be performed.
  Interventions: Procedure: "Distal Flap Reduction" Group
- "Only Exodontia" Group (Active Comparator): Exodontia of the 3rd molar will be performed following the different steps in the simple exodontic technique without performing any other surgical procedure.
  Interventions: Procedure: "Only Exodontia" Group

INTERVENTIONS:
Procedure: "Distal Flap Reduction" Group — A surgical procedure consisting of a tissue reduction flap distal to the second molar prior to the extraction of the third molar will be performed.
  Arms: "Distal Reduction Flap" Group
Procedure: "Only Exodontia" Group — Third molar exodontia without associated surgery.
  Arms: "Only Exodontia" Group

SUMMARY:
On many occasions, clinicians find situations in which they have to perform extractions of erupted or semi-erupted third molars or wisdom teeth where there are pre-existing periodontal pockets distal to the second molars, caused by a bone defect due to periodontal disease or due to malposition of the wisdom tooth concerning the second molar.

After the extraction of an erupted or semi-included third molar, and as a consequence of factors related to dental malposition or bone defects caused by periodontal disease, periodontal pockets can arise on the distal surface of the second molar.

When such exodontia is performed conventionally without raising a flap or applying any suturing technique in which there is a primary closure of the wound, there is a greater probability of persistence of periodontal pockets; and, in the worst case, they may increase after healing and closure of the alveolus. The consequence would be the formation of an enlarged and unattached tissue on the distal aspect of the second molar.

The fact that periodontal pockets persist acts as an unfavorable prognostic factor. The predictive power of subsequent periodontal destruction increases since these are areas where bacteria will continue to accumulate (etiological factor of periodontal disease), and where the patient will not be able to access for their elimination and control. This is why a surgical technique called "distal wedge" has been proposed to eliminate these pockets.

To avoid this second surgical procedure, we propose a procedure immediately after the conventional exodontic technique; where after performing a small gingivectomy and lifting a mucoperiosteal flap based on periodontal respective surgery concepts, primary closure of the alveolus and repositioning of the flaps at the level of the bone crest is achieved, eliminating these pre-existing pockets. This requires the existence of sufficient keratinized gingiva to maintain a band of at least 2 mm of keratinized tissue after the gingivectomy, thus ensuring a correct adherent tissue that provides sealing and proper maintenance of the periodontal tissues around the tooth. The proposed technique has been termed a "distal reduction flap" (DRF).

DETAILED DESCRIPTION:
The study population will be the patients of the University Clinic of the Rey Juan Carlos University of Madrid.

A non-probabilistic selection method will be used in the Master's Degree in Periodontology and Osseointegration and the Integrated Adult Clinical Dentistry course, for those patients who meet the inclusion criteria for the study.

Patients will be assigned to the experimental and control groups by probabilistic methods using a table of random numbers.

Variables:

Independent Variable: Surgical technique. In the experimental group, the Distal Reduction Flap (DRF) technique and primary wound closure will be used. In the control group, the conventional exodontic technique and secondary wound closure will be used.

Dependent variables. The reduction of probing depth at 6 weeks (RPS6) and 18 weeks (RPS18) will be evaluated. Modifying variables: The contribution of the following socioeconomic variables will be assessed:

Sex (male, female) Age (years) Systemic Diseases (Yes, No) Medication (Specify which) Tobacco (Yes, No) Mechanical Dental Plaque Control (Manual Brushing, Electric Brushing, or both) Chemical Dental Plaque Control (Yes, No)

The sequence of work:

T.0: A first consultation "Interview" will be carried out in which the nature of the study will be explained to the patient. A check will be made to see if the patient meets the inclusion criteria to take part in the study.

Periodontal probing with a Hu-Friedy® CP15 probe with 1 mm markings with a range of 0 to 15 mm. There will be a periodontal pocket distal to the second molars (probing depth equal to or greater than 4 mm).

2. The patient must be periodontally stable: Periodontal probing equal to or less than 4 mm and with bleeding on probing (BOP) index less than 25%.

3. Measure the amount of keratinized gingiva on vestibular and lingual/palatal second molars with a Hu-Friedy® CP15 periodontal probe, measuring the distance between the gingival margin and the amelo-cement line. There will be a minimum of 3 mm, to make a 1 mm buckle and keep at least a 2 mm band remaining.

4. Photographic records with Nikon®D5200 digital SLR camera body, with Nikon® compatible Sigma® 50 mm macro lens, Meke® ring flash, side mirror, and lip retractors.

T.1: On the day of surgery the working procedure will consist of:

* Anesthetic technique will be performed with infiltrative injection if it is in the upper jaw for blockade of the Posterior Alveolar Nerve and Palatine Nerve Major and Minor, and if it is in the lower jaw, regional injection will be performed for blockade of the Inferior Dental Nerve, Lingual Nerve and infiltrative for blockade of the Buccal Nerve. With Articaine 4% with epinephrine at 1:100.000. Ultracain ® (Normon® Laboratories, Madrid, Spain).
* The intervention will be performed according to the assigned randomization.

T.2: A review will be performed after 14 days and a photographic record will be taken, together with suture removal in the case of the study group. Post-operative discomfort perceived by the patient during the 3 days following the intervention will be recorded using V.A.E.

T.3: A review will be carried out 6 weeks after the intervention, where in addition to a photographic record, periodontal probing will be repeated with a Hu-Friedy® CP15 probe in the distal part of the 2nd molar. The reduction, persistence, or increase of the pre-existing periodontal pocket will be assessed.

T.4: A check-up will be performed at 12 weeks (18 weeks after the intervention). A new periodontal probing with a Hu-Friedy® CP15 probe in the distal part of the 2nd molar and a new photographic record will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require third molar extraction and who have periodontal pockets distal to the adjacent second molars.
* In the second molars there should be enough keratinized gingiva to allow for a buccal and/or lingual-palatal buckle (minimum residual band of 2 mm).
* Patients of either sex.
* Patients over 18 years old.
* Healthy patients or in a controlled periodontal situation (previously treated with basic periodontal therapy with scaling and root planing with probing depths of less than 4 mm and bleeding index at probing <25%).
* In the case of pharmacologically treated patients, they should be properly controlled and request prior consultation to evaluate pharmacological treatments that may lead to hematological alterations.

Exclusion Criteria:

* Patients with uncontrolled pathologies or systemic conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 6 and 18 weeks
  changes in probing depth

SECONDARY OUTCOMES:
Post-operative pain | 3 days
  A Visual Analog Scale (VAS) will be made to record the patient's assessment of the discomfort. The values of the scale will range from 1 to 10, with 1 being the score with the least pain and 10 being the score with the most postoperative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Francisco López Sánchez, MD, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Clinica Universitaria Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson RE. The distal wedge operation. Periodontics. 1966 Sep-Oct;4(5):256-64. No abstract available. PMID 5223126
- [Background] Matuliene G, Pjetursson BE, Salvi GE, Schmidlin K, Bragger U, Zwahlen M, Lang NP. Influence of residual pockets on progression of periodontitis and tooth loss: results after 11 years of maintenance. J Clin Periodontol. 2008 Aug;35(8):685-95. doi: 10.1111/j.1600-051X.2008.01245.x. Epub 2008 Jul 23. PMID 18549447
- [Background] Lindhe J, Socransky SS, Nyman S, Haffajee A, Westfelt E. "Critical probing depths" in periodontal therapy. J Clin Periodontol. 1982 Jul;9(4):323-36. doi: 10.1111/j.1600-051x.1982.tb02099.x. PMID 6764782
- [Background] Lang NP, Loe H. The relationship between the width of keratinized gingiva and gingival health. J Periodontol. 1972 Oct;43(10):623-7. doi: 10.1902/jop.1972.43.10.623. No abstract available. PMID 4507712
- [Background] Miyasato M, Crigger M, Egelberg J. Gingival condition in areas of minimal and appreciable width of keratinized gingiva. J Clin Periodontol. 1977 Aug;4(3):200-9. doi: 10.1111/j.1600-051x.1977.tb02273.x. PMID 330574
- [Background] Stetler KJ, Bissada NF. Significance of the width of keratinized gingiva on the periodontal status of teeth with submarginal restorations. J Periodontol. 1987 Oct;58(10):696-700. doi: 10.1902/jop.1987.58.10.696. PMID 2444693
- [Background] Claffey N, Nylund K, Kiger R, Garrett S, Egelberg J. Diagnostic predictability of scores of plaque, bleeding, suppuration and probing depth for probing attachment loss. 3 1/2 years of observation following initial periodontal therapy. J Clin Periodontol. 1990 Feb;17(2):108-14. doi: 10.1111/j.1600-051x.1990.tb01071.x. PMID 2406292
- [Background] Heitz-Mayfield LJ, Lang NP. Surgical and nonsurgical periodontal therapy. Learned and unlearned concepts. Periodontol 2000. 2013 Jun;62(1):218-31. doi: 10.1111/prd.12008. PMID 23574468